CLINICAL TRIAL: NCT05206903
Title: Emotional and Physical Health Status of Adults in Pandemia
Brief Title: Emotional and Physical Health Status of Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşe Ünal, PT., PhD., Pamukkale University
Other Study IDs: 21.01.2022/pandemia.awareness
Record Dates: First submitted 2022-01-21; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Pandemic, COVID-19; Adult ALL
Keywords: Pandemia awareness; General fatique; Quality of life; Sleep quality; Bodily pain; Status of physical activity
MeSH Terms: conditions — COVID-19; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sleep Initiation and Maintenance Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Questionnaires about pandemia process

SUMMARY:
To investigate the comparison of differences between emotional and physical health status of adults in COVID-19 isolation period and controlled normalization period.

ELIGIBILITY:
Inclusion Criteria:

* To speak Turkish
* Living in Turkey in pandemic process.
* Between the ages of 20-60 years.
* No communication problems.
* Being volunteer to participate in study.

Exclusion Criteria:

* Having communication problems.
* Not completion the assessments.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults between the ages of 20-60 years.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-06-10 (Estimated)

PRIMARY OUTCOMES:
Pandemic Awareness Scale | 1 minute
  To investigate the public pandemia awareness
Chalder Fatigue Scale | 2 minutes
  A self-report scale which is used to assess perceived fatique.
Pittsburgh Sleep Quality Index | 3 minutes
  A self-report scale
EQ-5D Health-Related Quality of Life Questionnaire | 1 minute
  This scale consists of 5 dimensions as mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Physical Activity Score | 1 minute
  The level of physical activity

IPD SHARING:
Plan to Share IPD: No